CLINICAL TRIAL: NCT04797442
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial to Evaluate the Effect of Akkermansia Muciniphila WST01 Strain in Patients With Type 2 Diabetes
Brief Title: Effect of Akkermansia Muciniphila WST01 Strain in Overweight or Obese Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, PHD, MD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WST001
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Obese; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: WST01 strain product
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: placebo powder

INTERVENTIONS:
Drug: WST01 strain product — orally given WST01 strain product, added onto lifestyle. The specific ingredients are the optimized Akkermansia muciniphila WST01 strain powder with maximum live bacteria of 5*10^10 CFU/g (1 g/pack, 3 packs QD, 20-30 min after breakfast)
  Arms: Experimental
Drug: placebo powder — orally given placebo powder (the specific ingrdients are the excipients of the WST01 strain powder), added onto lifestyle. (3 packs of placebo powder QD, 20-30 min after breakfast)
  Arms: Placebo comparator

SUMMARY:
The purpose of this study is to conduct a randomized, double-blinded, placebo-controlled, multicenter clinical trial, evaluating the glucose-lowering and weight-loss effects of Akkermansia muciniphila WST01 strain in overweight or obese patients with Type 2 Diabetes.

DETAILED DESCRIPTION:
In the present study, about 60 overweight/obese and drug naïve type 2 diabetes patients will be enrolled from multiple centers in China. After screening, eligible subjects will be randomized (1:1) into two groups, taking either Akkermansia muciniphila WST01 strain product or placebo product for 12 weeks.

Blood, feces and urine samples will be collected before and after treatment. Metabolic parameters including waist and hip circumference, area of visceral and subcutaneous fat, glycosylated hemoglobin (HbA1c), fasting plasma glucose (FPG), postprandial plasma glucose (PPG), insulin, glucagon-like peptide 1 (GLP-1), inflammation factors and lipid levels will be measured. Furthermore, the change of gut microbiota and metabolites will be evaluated too.

The primary objective is to determine whether Akkermansia muciniphila WST01 strain has a positive effect in patients with Type 2 Diabetes. The secondary objective is to explore the effect of Akkermansia muciniphila WST01 strain on safety, intestinal flora, insulin sensitivity, and other metabolic indicators and metabolites in the patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects with type 2 diabetes mellitus;
2. Age 18-60 years;
3. Overweight / obesity (24.0 ≤ BMI ≤ 40.0 kg/m2)；
4. Subjects with or without other obesity related metabolic complications (hypertension, dyslipidemia, hyperuricemia, etc.);
5. Subjects with screening HbA1c ≥ 7.0% and ≤ 10.0%, and the fasting blood glucose ≥ 7.0 mmol/l and ≤ 13.3 mmol/l；
6. Subjects who are not taking any medications to control blood glucose;
7. Subjects control blood glucose only by lifestyle intervention (diet and exercise) for at least 2 months before the screening period;
8. Subjects understand the nature, significance, potential benefits, inconvenience, and risks of the study before it starts；
9. Subjects fully understand the study produces and voluntarily sign the informed consent form.

Main Exclusion Criteria:

1. Subjects with a history of taking hypoglycemic drugs;
2. Subjects who are pregnant or in lactation;
3. Subjects with type 1 diabetes, single gene mutation diabetes, diabetes due to pancreatic injury or other secondary diabetes (such as Cushing's syndrome, thyroid dysfunction or acromegaly, etc.);
4. Subjects who were or are using oral hypoglycemic agents or insulin or incretin to control diabetes;
5. Subjects with liver and kidney dysfunction (alanine transaminase(ALT) / aspartate aminotransferase(AST)≥2.5×the upper limit of normal(ULN) set by the hospital, serum creatinine>1×ULN set by the hospital, or eGFR<60mL/min/1.73m2);
6. Surgery with serious cardiovascular and cerebrovascular diseases (such as heart failure, myocardial infarction, cerebral infarction, acute myocarditis, severe arrhythmia, patients receiving interventional therapy, etc.) or stage III hypertension (systolic blood pressure cannot be controlled below 160 mmHg with three antihypertensive drugs);
7. Subjects with acute diabetic complications such as diabetic ketoacidosis or diabetic hyperosmolar coma in the past 3 months;
8. Subjects with a medical history of malignant tumor (except local skin basal cell carcinoma) in the past 5 years;
9. Subjects with a medical history of intestine, or other digestive tract surgery (such as cholecystectomy) within one year, or other non-gastrointestinal surgery within 6 months;
10. Any condition that in the judgement of the investigator precludes participation.

Details please see the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  change of body weight from baseline
Fasting plasma glucose levels | 12 weeks
  change of fasting plasma glucose from baseline

SECONDARY OUTCOMES:
Gut microbiome | 12 weeks
  including fecal intestinal flora metagenome
Glycated haemoglobin (HbA1c) | 12 weeks
2-hour post-prandial plasma glucose levels | 12 weeks
Fasting serum insulin levels | 12 weeks
2-hour post-prandial serum insulin levels | 12 weeks
Fasting glucagon-like peptide-1 (GLP-1) levels | 12 weeks
2-hour post-prandial GLP-1 levels | 12 weeks
Serum triglycerides | 12 weeks
Serum total cholesterol | 12 weeks
Serum LDL-c | 12 weeks
Serum HDL-c | 12 weeks
Area of visceral and subcutaneous fat | 12 weeks
Waist and hip circumference | 12 weeks
Energy expenditure | 12 weeks
  using metabolic chamber to measure energy expenditure
Blood metabolomics profile measurement | 12 weeks
  In aid of LC/MS and GC/MS technique, etc, we will measure the metabolomics molecular profile in blood samples before and after treatment. The metabolomics measurement will help to detect the profile of all kinds of bile acid species, lipids species and amino acid species, etc. The composition change of all these biological molecular induced by the treatment is our major interest rather than single molecular quantification.
Inflammation markers | 12 weeks
  including hs-CRP, TNF-alfa, IL-6, and IL-8, etc
Systolic and diastolic blood pressure | 12 weeks
  Safety outcomes
Body temperature | 12 weeks
  Safety outcomes
Pulse rate | 12 weeks
  Safety outcomes
White blood cell (WBC) count | 12 weeks
  Safety outcomes
Red blood cell (RBC) count | 12 weeks
  Safety outcomes
Hemoglobin levels | 12 weeks
  Safety outcomes
Platelet count | 12 weeks
  Safety outcomes
Hepatic function | 12 weeks
  including alanine aminotransferase, aspartate aminotransferase，ɣ-glutamyltransferase, and alkaline phosphatase
Renal function | 12 weeks
  including serum urea nitrogen, serum creatinine, and serum urinary acid
Adverse events | 12 weeks
  Safety outcomes
Fasting serum C peptide levels | 12 weeks
2-hour post-prandial serum C peptide levels | 12 weeks
Lean mass | 12 weeks
  using DEXA scan to measure lean mass
Fat mass | 12 weeks
  using DEXA scan to measure fat mass

CONTACTS AND LOCATIONS:
Locations (1):
- Dep.endocrinology of Shanghai Ruijin Hospital, Shanghai Jiaotong university school of medcine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Y, Liu R, Chen Y, Cao Z, Liu C, Bao R, Wang Y, Huang S, Pan S, Qin L, Wang J, Ning G, Wang W. Akkermansia muciniphila supplementation in patients with overweight/obese type 2 diabetes: Efficacy depends on its baseline levels in the gut. Cell Metab. 2025 Mar 4;37(3):592-605.e6. doi: 10.1016/j.cmet.2024.12.010. Epub 2025 Jan 28. PMID 39879980